CLINICAL TRIAL: NCT06090110
Title: Clinical Efficacy of Transcutaneous Auricular Vagal Nerve Stimulation in Irritable Bowel Syndrome and the Potential Predictive Role for the Vagal-Autonomic Neurosignature
Brief Title: Vagal Nerve Stimulation in Irritable Bowel Syndrome
Acronym: RESILIENCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL84720.068.23
Record Dates: First submitted 2023-10-03; First posted 2023-10-19 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Irritable Bowel Syndrome
Keywords: vagal nerve stimulation
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): transcutaneous auricular vagal nerve stimulation, for 8 weeks at least one hour a day
  Interventions: Device: Vagal Nerve Stimulation
- placebo (Placebo Comparator): sham stimulation with a non-conducting electrode, for 8 weeks at least one hour a day
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Vagal Nerve Stimulation — Transcutaneous Auricular Vagal Nerve Stimulation
  Arms: Intervention
Device: Sham stimulation — Sham stimulation with a non-conduction electrode
  Arms: placebo

SUMMARY:
This randomized control trial aims to evaluate the effect of transcutaneous auricular vagal nerve stimulation in patients with irritable bowel syndrome. The intervention will be 8 weeks of treatment with a vagal nerve stimulator. The main objectives are:

* To evaluate the clinical response, defined as a decrease of at least 50 points on the IBS-SSS questionnaire, of the treatment.
* To ascertain whether the autonomic-vagal neurosignature, derived from pre-treatment registration of symptom profiles, autonomic responses and imaging of neuronal activity as a reaction to stress is able to predict therapeutic response to tVNS accurately.
* To evaluate the effect of treatment on quality of life
* To evaluate the effect of treatment on depression
* To evaluate the effect of treatment on anxiety Participants will be asked to wear a wearable (Fitbit) and fill out a daily questionnaire for one week. Thereafter, a functional brain MRI will be performed.

In the intervention group patients will receive transcutaneous nerve stimulation for 8-weeks at home. The comparison group will receive the same device but with a non-conducting electrode.

Patients fill out weekly questionnaires during the treatment period and at follow-up moments 3 and 6 months after finishing the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of IBS according to Rome IV criteria (3), as follows:
* Recurrent abdominal pain, on average, at least 1 day per week in the last 3 months, associated with 2 or more of the following criteria:
* Related to defecation.
* Associated with a change in stool frequency.
* Associated with a change in stool from (appearance).
* Criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis.
* Age between 18 and 75 years;
* Ability to understand and speak the Dutch language.
* Ability to understand how to utilize the ESM application.

Exclusion Criteria:

* A history of abdominal surgery, except for uncomplicated appendectomy, laparoscopic cholecystectomy and hysterectomy is present or otherwise based on the principal investigator's judgement.
* Presence of metallic prostheses, pacemakers, metal clips on blood vessels, metal parts in the eye, an intrauterine device (with the exception of the Mirena IUD), metal braces, facial tattoos and/or metal objects.
* History of major head trauma or head/brain surgery
* History of claustrophobia
* Pregnancy, lactation, intention to become pregnant during the study period
* Students and employees of Maastricht University are not precluded from participation, unless they have a direct personal, professional or hierarchical position with regards to any of the study team members or their department.
* If the subject has a cardiac arrhythmia, the attending physician will be consulted before participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Clinical meaningful decrease in severity of GI-symptoms | at the end of the 8 week treatment period
  Measuring IBS-SSS, defined as a decrease of at least 50 points

SECONDARY OUTCOMES:
Predictive value of neuro-signature | at the end of the 8 week treatment period
  The value of the multimodal neuro-signature in the prediction of clinical response to tVNS in IBS-patients.
adverse events | at the end of the 8 week treatment period
  Number and severity of adverse events
Anxiety/depression | at the end of the 8 week treatment period
  Symptoms of anxiety and depression measured using PHQ-9 and GAD-7
Cost-effectiveness | at follow up moment 2 (6 months after 8 week treatment period)
  Direct and indirect costs made during the treatment period
Time the device was used | at the end of the 8 week treatment period
  The amount of time patients used the tVNS device

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Keszthelyi, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands